CLINICAL TRIAL: NCT05522920
Title: Non-invasive Spinal Cord Stimulation Combined With Activity-based Therapy in Chronic Complete High Level Spinal Cord Injury
Brief Title: Spinal Stimulation for Chronic Complete Tetraplegia
Acronym: Complete TESCS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: International Spinal Research Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN20NE064
Record Dates: First submitted 2022-08-25; First posted 2022-08-31 (Actual); Last update posted 2022-08-31 (Actual); Status verified 2022-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Therapeutics; Spinal Cord Stimulation

STUDY DESIGN:
Intervention Model Description: All participants will receive study intervention
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Therapy (Experimental): Conventional physical therapy will be used with and without spinal cord stimulation to investigate improvement of upper limb function.
  Interventions: Other: Therapy with and without spinal cord stimulation

INTERVENTIONS:
Other: Therapy with and without spinal cord stimulation — Conventional therapy only will be followed with conventional therapy combined with electrical spinal cord stimulation.

SUMMARY:
The purpose of this study is investigate the acceptability and effectiveness of transcutaneous spinal cord stimulation in people with complete high level spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give informed consent for participation in the study
* Aged ≥18 years
* Injury level C3-C7, American Spinal Cord injury Association Impairment Scale (ASIA) A
* ≥1 year post-injury
* Medically stable, cognitively intact, and able to breathe independently
* Able to attend all sessions two or three times per week, for 2 h sessions and assessments

Exclusion Criteria:

* Any implanted active metallic device including, but not limited to neurostimulators, cochlear implants, pacemakers, implantable defibrillators, or drug delivery pumps
* Possible, suspected, or confirmed pregnancy and/or lactation
* Recent history or fracture, contractures or pressure sore, deep vein thrombosis (DVT) or urinary tract, or other infection that may interfere with the intervention and training
* History of epilepsy and/or seizures
* Severe spasticity which has been unstable over the 3 months prior to enrolment and is not expected to change and/or taking varying doses of anti-spasticity medications which could not be tapered to a stable dose and are not expected to change
* Botulinum toxin injections within 6 months of participation
* Non-injury related neurological impairment
* Clinically significant severe depression in spite of treatment
* Cardiovascular disease
* Autonomic dysreflexia that is severe, ongoing, and has required medical treatment within the past month
* Skin conditions or allergies that may affect electrode placement
* Do not understand English
* Received a stem cell treatment or other treatment that could possibly promote or attenuate neuroplastic changes in spinal or cortical function, within ≥2 years of enrolment; beyond this period, they may be included, provided the treatment was conducted in an accredited facility with proper ethics and regulatory approval.
* Involved in any other study involving stimulation of the spinal cord within 6 months of enrolment
* Information regarding recent rehabilitation or exercise programmes that participants may currently be engaged in will be discussed with clinical staff and fully documented for each participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Acceptance | 26 weeks at the end of intervention
  Whether the treatment protocol is acceptable by people with complete tetraplegia. This will be assessed using semi structured interview results of which will be analysed qualitatively to determine the number of participants who would use the therapy on an ongoing basis.

SECONDARY OUTCOMES:
Clinical effectiveness of spinal cord stimulation using GRASSP tool | 26 and 38 weeks, at the end of intervention and at follow up respectively
  Effectiveness of spinal cord stimulation in inducing changes in functional outcome. This will be assessed using the Graded and Redefined Assessment of Strength, Sensibility, and Prehension (GRASSP tool). The unit is based on the GRASSP measurement scale.
Neurophysiological change | 26 and 38 weeks, at the end of intervention and at follow up respectively
  Effectiveness of spinal cord stimulation in inducing changes in Neurophysiological equivalence of volitional movement. This will be assessed using changes in amplitude in mV of transcranial magnetic stimulation.
Sensation | 26 weeks at the end of intervention
  Change in sensation due to the intervention. This will be assessed using change the sensory score of the International Standards for Neurological classification of SCI (ISNCSCI)
Spasticity | 26 weeks at the end of intervention
  Changes in upper limb muscle tone using change in the Modified Ashworth Scale.
Autonomic function | 26 weeks at the end of intervention
  Changes in autonomic function will be assessed using changes in the AUTONOMIC STANDARDS ASSESSMENT FORM of the International Spinal Cord Injury Data Set.
Change in perceived health status | 26 weeks at the end of intervention
  The effect of the study on perceived health status of the participants will be assessed using QUALITY OF LIFE BASIC DATA SET of the International Spinal Cord Injury Data Set.

CONTACTS AND LOCATIONS:
Overall Officials: Mariel Purcell, Consultant, Study Director — NHS Greater Glasgow and Clyde

IPD SHARING:
Plan to Share IPD: Undecided
The is no plan yet to share individual participant data.

REFERENCES:
- [Derived] McNicol EL, Osuagwu B, Purcell M, McCaughey EJ, Lincoln C, Cope L, Vuckovic A. Neurophysiological Effect of Transcutaneous Electrical Spinal Cord Stimulation in Chronic Complete Spinal Cord Injury. Artif Organs. 2025 Jun 30. doi: 10.1111/aor.15050. Online ahead of print. PMID 40583777